CLINICAL TRIAL: NCT05445297
Title: Prospective Randomized Study Comparing the Efficacy and Safety of Refralon and Amiodarone in Cardioversion in Patients With Paroxysmal Atrial Fibrillation and Flutter
Brief Title: Refralon Versus Amiodarone for Cardioversion of Paroxysmal Fibrillation and Atrial Flutter
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JCBY-2021-0007-275
Record Dates: First submitted 2022-06-27; First posted 2022-07-06 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation Paroxysmal
Keywords: atrial fibrillation and flutter; paroxysmal atrial fibrillation and flutter; cardioversion AF; Amiodarone; Refralon; Niferidil; new antiarrhythmic drug; new Russian antiarrhythmic drug refralon
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amiodarone group (Other)
  Interventions: Drug: Pharmacological cardioversion with Amiodarone
- Refralon group (Other)
  Interventions: Drug: Pharmacological cardioversion with Refralon

INTERVENTIONS:
Drug: Pharmacological cardioversion with Amiodarone — Patients in this group will receive intravenous amiodarone according to the following scheme:
  1. administration of 5 mg/kg body weight of amiodarone diluted in 250 ml of 5% glucose solution intravenously for 20-60 minutes, depending on the tolerability of the drug.
  2. if there is no effect (recovery of SR did not occur within 60 minutes from the start of the drug administration), continue the infusion of amiodarone intravenously at a dose of 100 mg/hour until a total dose of 1200 mg is reached.
  Other Names: Amiodarone
  Arms: Amiodarone group
Drug: Pharmacological cardioversion with Refralon — Patients in this group will receive intravenous refralon according to the following scheme:
  1. the introduction of a 0.1% solution of refralon at a dose of 5 μg per 1 kg of body weight, diluted in 20 ml of saline intravenously for 2-3 minutes;
  2. in the absence of effect (SR recovery did not occur), after 15 minutes, repeated intravenous administration of a 0.1% solution of refralon at a dose of 5 μg per 1 kg of body weight (total dose of the drug 10 μg / kg of body weight);
  3. in the absence of effect (SR recovery did not occur), after 15 minutes, the next intravenous injection of a 0.1% solution of refralon at a dose of 10 μg per 1 kg of body weight (total dose of the drug 20 μg / kg of body weight);
  4. in the absence of effect (recovery of SR did not occur), after 15 minutes, repeated intravenous administration of a 0.1% solution of refralon at a dose of 10 μg per 1 kg of body weight. Thus, the maximum total dose of the drug will be 30 μg/kg of body weight.
  Other Names: Refralon
  Arms: Refralon group

SUMMARY:
Patients hospitalized with paroxysmal atrial fibrillation and flutter to restore sinus rhythm will be randomized into two groups: one will be cardioversion with refralon and the other with amiodarone

DETAILED DESCRIPTION:
Atrial fibrillation (AF) and flutter (AFL) are the most common types of arrhythmia in clinical practice. Both electrical and medical cardioversion can be used to restore sinus rhythm. Currently, the most studied and commonly used drug for pharmacological cardioversion of paroxysms of AF/AFL is amiodarone, which belongs to class III antiarrhythmic drugs. The highest recovery rates of sinus rhythm (SR) (>90%) are achieved with intravenous administration of amiodarone at a dose of more than 1500 mg / day or up to a maximum of 3000 mg / day. However, most commonly, amiodarone is used at a standard dose of 5 mg/kg body weight, with an efficacy of 34-69%. In 2014, a new Russian class III antiarrhythmic drug, Refralon, was registered. In 2020, the drug was included in the National Clinical Guidelines "Atrial Fibrillation and Flutter", approved by the Ministry of Health of the Russian Federation. When using refralon in doses from 10 to 30 μg/kg, SR recovery was noted in 91.6% of patients with persistent AF/AFL in 50% of patients SR restored within 15 minutes from the start of the drug administration.

Randomized trials comparing the efficacy and safety of refralon with other antiarrhythmic drugs have not been conducted. It is extremely important to directly compare the efficacy and safety of these two drugs in patients with paroxysmal AF in a prospective randomized study.

ELIGIBILITY:
Inclusion Criteria:

1. Paroxysmal form of AF/AFL;
2. Indications for SR recovery

Exclusion Criteria:

1. Arrhythmogenic effect of refralon, amiodarone and other antiarrhythmic drugs in history;
2. Chronic kidney disease with a decrease in glomerular filtration rate less than 30 ml / min / 1.73 m2;
3. Chronic heart failure (functional class IV);
4. Atrioventricular blockade of 2-3 degrees (with the exception of patients with an implanted pacemaker);
5. Dysfunction of the sinoatrial node (with the exception of patients with an implanted pacemaker);
6. Bradysystolic atrial fibrillation (heart rate <50 beats/min);
7. Duration of the QT interval >440 ms;
8. Hemodynamic instability requiring emergency cardioversion;
9. Contraindications to anticoagulant therapy;
10. Thyrotoxicosis or decompensated hypothyroidism;
11. Uncorrected electrolyte disturbances at the time of cardioversion (potassium level less than 3.5 mmol/l);
12. Pregnancy and breastfeeding period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Restoration of sinus rhythm | 1 hour
  Restoration of SR within 1 hour from the start of drug administration (refralon/amiodarone).
Restoration of sinus rhythm | 24 hours
  Restoration of SR within 24 hour from the start of drug administration (refralon/amiodarone).
Number of patients who recovered sinus rhythm after the minimum dose of refralon. | 24 hours
  Number of patients who recovered SR when using refralon at a dose of 5 µg/kg.
Sinus rhythm recovery time | 24 hours
  The time elapsed from the start of drug administration to recovery of SR
Recurrent AF/AFL after successful cardioversion | 24 hours
  Absence of sustained (more than 30 seconds) recurrences of AF/AFL within 24 hours after successful cardioversion;
Ventricular arrhythmogenic effect | 24 hours
  Registration of sustained and nonsustained (3 or more QRS) ventricular tachycardia or ventricular fibrillation after administration of drug (refralon/amiodarone)
Increased QT interval (more than 500 ms) | 24 hours
  The number of patients who have an increase in the QT interval (more than 500 ms) and the time during which the duration of the QT interval exceeded 500 ms.
Bradyarrhythmias (pauses and bradycardia) | 24 hours
  Decrease in heart rate to less than 50bpm after administration of drug (refralon/amiodarone) during AF or after restoration of SR - the minimum heart rate, the duration of the maximum recorded pause and the time during which the heart rate was less than 50bpm will be recorded
Arterial hypotension | 24 hours
  Decrease in blood pressure by more than 20 mm Hg from the initial value(if asymptomatic) after administration of drug (refralon/amiodarone) or by more than 10 mm Hg (if symptomatic)
Any clinical manifestations | 24 hours
  The appearance of any clinical manifestations after administration of drug (refralon/amiodarone) that are interpreted by the doctors of the intensive care unit as a worsening of patient's clinical status.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Budgetary Institution NATIONAL MEDICAL RESEARCH CENTRE OF CARDIOLOGY NAMED AFTER ACADEMICIAN E.I.CHAZOV. of the Ministry of Health of the Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No